CLINICAL TRIAL: NCT04546737
Title: Study of Morphological, Spectral and Metabolic Manifestations of Neurological Complications in Covid-19 Patients
Acronym: NSpectroCovid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2020_843_0087
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Neurological Manifestations; Brain Damage
Keywords: Covid19; Neurological Manifestations; MRI and NMR spectroscopy; Radiological semiology; Spectral profile; Brain Damage
MeSH Terms: conditions — COVID-19; Neurologic Manifestations; Brain Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Magnetic Resonance Spectroscopy (MRS). — This is a Nuclear Magnetic Resonance (NMR) technique which can detect the NMR signal allowing to measure under curves areas, amplitudes, ratios and concentrations of various metabolites contained in a biological tissue, in addition to water and lipids. This offers the possibility, in addition to the contribution of MRI imaging, to better characterize pathological processes (inflammatory, infectious, etc.) through spectral and metabolic changes that can be quantitatively evaluated. Spectroscopic measurements will be carried out with a mono-voxel spectroscopy using a PRESS [Point RESolved Spectroscopy] sequence with a short Echo Time (TE) of 35 ms, an intermediate TE of 144 ms and a long TE of 288 ms.

SUMMARY:
Viral pandemics, such as HIV and SARS-Cov-V1, have shown that they can lead to acute and / or delayed neurological complications. At the actual context of the pandemic Coronavirus disease 2019 (COVID-19), neurological manifestations seem to be confirmed since in 85% of COVID-19 patients, present neurological symptoms, including anosmia, ageusia, periorbital pain, dizziness, fatigue, even moderate headache, moderate memory and/or behavioral disorders.

However, these neurological manifestations are not well studied and their radiological features are not well described. It is therefore important to assess these potential neurological complications in COVID-19 patients. To the investigator knowledge, there is no previous study in the literature describing spectral brain changes in COVID + patients. Thus, the goal of this work is to describe the radiological semiology using MRI and particularly Magnetic Resonance Spectroscopic (MRS) biomarkers in the evaluation of acute and / or delayed brain damage in COVID + patients presenting a neurological manifestations that are initially related to the cranial nerves damage.

ELIGIBILITY:
Inclusion Criteria:

* Major COVID-19 patient (≥18 years old)
* COVID-19 patient presenting at least one the neurological manifestations:

anosmia, ageusia, periorbital pain, dizziness, fatigue, moderate headache, moderate memory and behavioral disorders.

* Patient who have signed an informed consent form for the study

Exclusion Criteria:

* Patient under guardianship or curators or under judicial protection
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Variation from baseline of MRI radiological semiology in COVID-19 patients | 9 months after patient inclusion
  The radiological semiology as described by MRI and particularly Magnetic Resonance Spectroscopic (MRS) biomarkers in the COVID-19 patients presenting neurological manifestations related initially to the cranial nerves damage.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No